CLINICAL TRIAL: NCT00676312
Title: A Partially-Blinded, Randomized, Placebo and Active Controlled, Ascending Single-Dose Crossover Phase I Study to Explore the Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Effects of PTH134 Formulated With Different Concentrations of 5-CNAC in Healthy Postmenopausal Women
Brief Title: Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Effect of PTH134 at Increasing Doses in Healthy Postmenopausal Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CPTH134A2101
Record Dates: First submitted 2008-05-08; First posted 2008-05-13 (Estimated); Last update posted 2008-12-11 (Estimated); Status verified 2008-12

CONDITIONS: Postmenopausal Osteoporosis
Keywords: Osteoporosis; parathyroid hormone; pharmacodynamic; pharmacokinetic
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Osteoporosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (1):
- 1 (Experimental): Cross-over treatment with increasing doses of PTH134, placebo and active comparator.
  Interventions: Drug: PTH134

INTERVENTIONS:
Drug: PTH134
  Other Names: teriparatid

SUMMARY:
This study is designed to investigate the safety and tolerability of PTH134 in healthy subjects and to assess the exposure from PTH134.

ELIGIBILITY:
Inclusion Criteria:

* Healthy postmenopausal female subjects, 40 to 70 years of age and in good health as determined by past medical history, physical examination, vital signs, electrocardiogram, and laboratory tests at screening
* Body mass index (BMI) within the range of 19 to 32.

Exclusion Criteria:

* Smokers who report cigarette use of >= 5 cigarettes per day.
* Use of any prescription drugs or over-the-counter (OTC) medication (vitamins, herbal supplements, dietary supplements) started within the last month prior to screening.
* Previous osteoporosis treatment
* History of drug or alcohol abuse within the 12 months prior to dosing or evidence of such abuse

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 40 Years to 70 Years | Sex: Female
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2008-05; Primary Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
•Safety and tolerability of ascending single doses of PTH134 over 24 hours as compared to baseline. •Pharmacokinetics after ascending single doses of PTH134, including comparison with reference drug Forteo 20 µg sc over 24 hours.

SECONDARY OUTCOMES:
•Assessment of PK from PTH134 formulations over 24 hours. •Assessment of the pharmacodynamic profile of serum ionized calcium, total serum calcium, bone biomarkers with reference drug Forteo 20 µg and placebo over 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharma AG, Basel, Principal Investigator — Novartis Pharma AG, Basel
Locations (1):
- Novartis Investigative site, Basel, Switzerland

REFERENCES:
- [Derived] Hammerle SP, Mindeholm L, Launonen A, Kiese B, Loeffler R, Harfst E, Azria M, Arnold M, John MR. The single dose pharmacokinetic profile of a novel oral human parathyroid hormone formulation in healthy postmenopausal women. Bone. 2012 Apr;50(4):965-73. doi: 10.1016/j.bone.2012.01.009. Epub 2012 Jan 25. PMID 22289659